CLINICAL TRIAL: NCT02939586
Title: A Cross-sectional, Randomised-controlled Study to Investigate the Effect of HDF vs HD in Sleep Apnoea
Brief Title: The Effect of Haemodialysis in Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Hunter Hospital (Other Government)
Collaborators: Newcastle University (Other); Hunter Medical Research Institute (Unknown)
Responsible Party: Principal Investigator, Ginger Chu, Clinical Nurse Consultant, John Hunter Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JohnHunterH
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Sleep Apnoea; Renal Failure; End Stage Kidney Disease; Sleep Disturbance; Sleep Disorders; Sleep
Keywords: Sleep, Sleep apnoea, Haemodialysis, Haemodiafiltration, end stage kidney disease
MeSH Terms: conditions — Sleep Apnea Syndromes; Renal Insufficiency; Kidney Failure, Chronic; Parasomnias; Sleep Wake Disorders | interventions — Dialysis

STUDY DESIGN:
Intervention Model Description: eligible participants from stage 1 screening will be invited to participate in stage 2 RCT. participants will be randomly assigned to either HD or HDF for 2 months, 1 month wash-our period and cross-over to the other treatment for another 2 months. The total trial period will be 5 months.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haemodialysis (Active Comparator): regular convectional haemodialysis 3times/weekly
  Interventions: Procedure: Haemodiafiltration post-dilution model
- Haemodiafiltration (Active Comparator): post-dilution haemodiafiltration
  Interventions: Procedure: Haemodialysis

INTERVENTIONS:
Procedure: Haemodiafiltration post-dilution model — Participants will be randomly assigned into either HD or HDF group. The participants will received the assigned treatment for 2 months, 1 month wash-out (HD) and cross-over to the other dialysis model- eg. HDF (2months) and switch to HD for 2 months, with 1 month washout period (using standard HD). Haemodialysis post-dilution model will be delivered using fresenius 5008 machine. Prescription for HDF post-dilution will be comparable to HD.
  Arms: Haemodialysis
Procedure: Haemodialysis — Participants will be randomly assigned into either HD or HDF group. The participants will received the assigned treatment for 2 months and cross-over to the other dialysis model- eg. HD (2months) and switch to HDF for 2 months, with 1 month washout period (using standard HD). Haemodialysis treatment will be delivered using fresenius 5008 machine. treatment time/parameters may vary depends on individual prescription.
  Arms: Haemodiafiltration

SUMMARY:
Sleep disturbance is a significant issue in people undergoing dialysis. More than 80% of haemodialysis patients complain of difficulty sleeping. Inadequate sleep can cause poor daytime function and increased risk of motor vehicle incidents.

One of the common reasons for sleep disturbance in dialysis patients is sleep apnoea. Sleep apnoea involves pauses in breathing that occur during sleep. Each pause can last only a few seconds or minutes. Severe sleep apnoea reduces oxygen supply and increases risk of heart attack and stroke, which are the leading causes of death in dialysis patients.

In this project, the investigators will examine how a change of dialysis treatment might improve sleep. This project will first identify patients at risk of sleep disturbance using surveys and a subsequent sleep study. The investigators will then test different dialysis models to see the effect of dialysis treatment on sleep apnoea. The aim is to find a dialysis model that works better for patients with sleep apnoea.

DETAILED DESCRIPTION:
Sleep Problem in Dialysis Patients Sleep apnoea is a significant issue in patients with end stage kidney disease. Evidence suggests that up to 80% of dialysis patients have sleep apnoea [1], yet the standard haemodialysis treatment does not improve the symptoms of sleep disturbance in most patients [2].

Sleep disturbance is specifically associated with poor quality of life (QoL) [4]; decreased mental and physical function, and adversely impact survival [5-7]. Recent data also suggest that the low oxygen state resulting from sleep apnoea can exaggerate the deterioration of kidney function and increase risk of high blood pressure, cardiovascular abnormality and overall death rates [8]. Despite the significance of sleep apnoea, it is acknowledged that there is insufficient evidence for clinicians to manage this common symptom burden in the dialysis population [9]; and patients who receive maintenance dialysis today still experience poor QoL and worse survival rates compared with most common cancer sufferers [10].

Knowledge Gap It is believed that the mechanism of sleep apnoea in dialysis patients are related to overactive chemoreceptors, which cause destabilisation of the respiratory drive and periodic breathing during the night [13]. Since the chemoreceptors can be triggered by inflammatory blood toxins, which accumulate in kidney failure [14], it is proposed that better clearance of these molecules can improve symptoms and outcomes of sleep apnoea. These molecules are poorly removed by standard haemodialysis [15] and are thought to cause the symptomatic effects of poor kidney function and inflammation, which are associated with poor sleep quality [16].

Better dialysis treatment may play an important role in the management of sleep apnoea. Previous studies have suggested that sleep apnoea may be improved by nocturnal dialysis; an intensive treatment which patients undergo at home, during sleep, for 8-10 hours every night. It provides better blood purification, compared with standard haemodialysis treatment. However, nocturnal dialysis is a home therapy which is not viable for the majority of haemodialysis patients who require care in a clinical setting. There is clearly a need to explore the effectiveness of dialysis treatment on sleep apnoea using a different dialysis model.

Modern dialysis technology, such as Haemodiafiltration (HDF), allows for better removal of toxic molecules such as beta 2 microglobulin (B2M) and C-Reactive protein (CRP), than standard haemodialysis treatment, and may offer the benefits of nocturnal dialysis to all dialysis patients. No one has examined the effect of HDF on sleep apnoea in haemodialysis patients, and the investigators will answer this question in this study.

Research Aims

1. To determine the prevalence of sleep apnoea in the local dialysis population using a validated questionnaire and sleep study. Although sleep apnoea is recognised as common in the dialysis population, there is a need to reproduce this data in the context of local dialysis services to accurately identify affected patients
2. To examine the effect of HDF compared conventional haemodialysis on health status and sleep quality in patients with sleep apnoea, using a randomised cross-over trial (RCT)
3. To determine if the clearance of middle-sized uraemic toxins improves symptoms of sleep apnoea. The middle-sized molecules to be assessed in this study include C-Reactive protein (CRP), beta 2-microglobulin (β2M), tumour necrosis factor alpha (TNF-α), interleukin 6 (IL-6), and interleukin 8 (IL-8), which are the serum inflammatory markers that are commonly found in patients with obstructive sleep apnoea.

ELIGIBILITY:
Inclusion criteria

* Individuals receiving maintenance haemodialysis under the care of Nephrology Department, John Hunter Hospital & Manning Base Hospital
* Have received dialysis for more than 3 months.
* Greater than 18 years of age
* Able to provide informed consent
* Satisfactory written and spoken English language skills
* AHI score between 15-29 or above 30 if the participant a. declines sleep apnoea treatment after discussing with their physician, b. would like to be involved in the trial whilst awaiting an appointment in the sleep clinic.

Exclusion criteria

* Acute dialysis or acutely unwell patients
* Home dialysis patients
* Unable to participate in the study in the opinion of the participant's primary Nephrologist or due to language barrier or cognitive impairment.
* Already on treatment for sleep-disordered breathing
* Woman who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Severity of Sleep Apnea measured by Apnea-hypopnea index | 18 months
  The Apnea-Hypopnea Index (AHI) score will be used to determine the severity of sleep apnea. The AHI will be obtained via an overnight sleep study. An AHI score of 5-14.9/hr is classified mild sleep apnea, 15-29.9/hr is moderate and above 30/hr is severe sleep apnea.

SECONDARY OUTCOMES:
Patient-reported sleep quality measured by PSQI | 18 months
  The subjective sleep quality will be measured by Pittsburgh Sleep Quality Index (PSQI). The PSQI is an effective tool to measure the quality and patterns of sleep, and to differentiate "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month period. A global sum of 5 or greater indicates "poor" sleep.
Patient-reported daytime sleepiness measured by ESS | 18 months
  The subjective sleep quality will also be measured by Epworth Sleepiness Scale (ESS). ESS is an eight-item survey that assesses an individual's level of daytime sleepiness. A score of greater than ten (out of 24) is considered to be indicative of abnormal sleepiness, and 16 or more as severe sleepiness
Overall quality of life measured by KDQoL-36 | 18 months
  Overall quality of life will be measured by Kidney Disease Quality of Life Instrument (KDQOL-36). This tool examines 20 variables which include renal specific measurements. The domains examined include physical and social functioning, physical and emotional role limitations, physical pain, mental health, vitality, general health perceptions plus the burden of kidney disease, and symptoms/problems commonly associated with kidney disease. The score of KDQoL-36 ranges from 0-100, and higher score indicates higher quality of life reported by patients.
The different concentration of inflammatory biomarkers (CRP, β2M, TNF-α, IL-6 and IL-8) during HDF period vs HD period, and the correlation to AHI, and overall sleep quality and quality of life. | 18 months
  Blood samples will be collected from eligible participants in stage 2, and analysed for inflammatory biomarkers concentration using Elisa kit.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa McDonald, PhD, Principal Investigator — Academic Clinician/University of Newcastle
Locations (2):
- Australia (2):
  - John Hunter Hospital, Newcastle, New South Wales
  - John Hunter Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No